CLINICAL TRIAL: NCT04722562
Title: Investigation of the Pharmacokinetics, Safety, and Tolerability of Vericiguat (BAY1021189) in Subjects With Hepatic Impairment (Classified as Child Pugh A or B) and in Age-, Weight-, and Gender-matched Healthy Subjects Following a Single Oral Dose in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: A Trial to Learn How Safe Vericiguat (BAY1021189) is and the Way the Body Absorbs, Distributes and Gets Rid of Vericiguat in Participants With Liver Disease and in Age-, Weight- and Gender-matched Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15840; 2014-001206-18 (EudraCT Number)
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child Pugh A (Experimental): Participants with mild hepatic impairment
  Interventions: Drug: Vericiguat (BAY1021189)
- Child Pugh B (Experimental): Participants with moderate hepatic impairment
  Interventions: Drug: Vericiguat (BAY1021189)
- Healthy participants (Experimental): Participants with normal hepatic function
  Interventions: Drug: Vericiguat (BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) — Oral single dose of 2.5 mg (2 x 1.25 mg immediate release tablet)

SUMMARY:
Vericiguat (BAY1021189) is under development to treat heart failure, a condition in in which the heart has trouble pumping blood through the body. Liver impairment which co-occurs in patients with heart failure is a common condition in which the liver is not removing the drugs from the blood as well as it should.

The goal of the study was to learn more about the safety of vericiguat (BAY1021189), how it was tolerated and the way the body absorbed, distributed and excreted the study dug given as a single oral dose of 2.5 mg tablet in participants with liver impairment and healthy participants matched for age-, gender-, and weight.

The participants stayed at the trial site for about 5 days. During this time, the doctors took blood and urine samples and checked the participants' health. About 7 after the participants took vericiguat (BAY1021189), the researchers checked the participants' health again and asked about any medical problems they had.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Aged between 18 and 79 years (inclusive) with body mass index 18 to 34 kg/m^2 (both inclusive)
* Women without childbearing potential; women of childbearing potential only if the pregnancy test was negative and a combination of condoms with a safe and highly effective

For subjects with hepatic impairment:

* Subjects with documented liver cirrhosis confirmed by histopathology, e.g., previous liver biopsy, laparoscopy, ultrasound, or fibroscan
* Subjects with hepatic impairment (Child Pugh A or B)
* Subjects with stable liver disease in the last 2 months

For healthy subjects:

* Mean age and body weight in the control group and in the two groups with hepatic impairment (Child Pugh A and B) should not vary by more than ± 10 years and ± 10 kg
* Gender matched

Exclusion Criteria:

For all subjects:

* Subjects with a medical disorder, condition, or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Medical history of Kock pouch (ileostomy after proctocolectomy)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known gastrointestinal (GI) disorders (eg stomach ulcers, duodenal ulcers, GI bleeding) or inflammatory bowel disease (eg Crohn's disease, ulcerative colitis)
* Febrile illness within 1 week prior to admission to study center
* Relevant diseases within the last 4 weeks prior to admission to study center
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Subjects with diagnosed malignancy within the past 5 years

For subjects with hepatic impairment:

* Severe cerebrovascular or cardiac disorders, e.g., myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association grade III or IV, severe arrhythmia requiring anti-arrhythmic treatment
* Evidence of hepatic encephalopathy related to chronic liver disease > grade 2 (exclusion by Number Connection Test (NCT))
* Subjects with percutaneous transluminal coronary angioplasty or coronary artery bypass graft less than 6 months prior to study drug administration
* History of bleeding within the past 3 months
* Thrombotic disorder
* Subjects with diabetes mellitus with a glycohemoglobin A1c (HbA1c) >10%
* Severe ascites of more than 6 L (estimated by ultrasound)
* Subjects with primary and secondary biliary cirrhosis
* Subjects with sclerosing cholangitis
* Failure of any other major organ system other than the liver
* Severe infection, malignancy, or psychosis, or any clinically significant illness within 4 weeks prior to study drug administration

For healthy subjects:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal
* Subjects with conspicuous findings in medical history or pre-study examination
* A history of relevant diseases of vital organs, the central nervous system, or other organs

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2015-01-21 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
AUC of vericiguat | Up to 96 hours
  Area under the concentration vs. time curve from zero to infinity after single dose administration
AUCu of vericiguat | Up to 96 hours
  AUC unbound
Cmax of vericiguat | Up to 96 hours
  Maximum observed drug concentration in measured matrix after single dose administration
Cmax,u of vericiguat | Up to 96 hours
  Cmax unbound

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Lübeck, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/